CLINICAL TRIAL: NCT06724692
Title: Acute Effects of Ultra-processed Versus Unprocessed Foods on Glucocorticoid Secretion in Healthy Individuals
Acronym: UltraCort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eleonora Seelig (Other)
Responsible Party: Sponsor-Investigator, Eleonora Seelig, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EKNZ 2024-01796
Record Dates: First submitted 2024-09-27; First posted 2024-12-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Glucocorticoids; Obesity and Overweight; Food Effect
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Randomized, monocentric, cross-over, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultra-processed breakfast (Active Comparator): During one study phase, subjects receive an ultra-processed breakfast
  Interventions: Other: Ultra-processed breakfast
- Low-processed breakfast (Active Comparator): During the other study phase, subjects receive a low-processed breakfast
  Interventions: Other: Low-processed breakfast

INTERVENTIONS:
Other: Ultra-processed breakfast — With this intervention, participants will consume ultra-processed foods
  Arms: Ultra-processed breakfast
Other: Low-processed breakfast — With this intervention, participants will consume low-processed foods
  Arms: Low-processed breakfast

SUMMARY:
The investigators aim to understand whether the acute cortisol response to food differs between differently processed foods.

In this monocentric, randomized, cross-over, open-label study, 20 healthy volunteers will receive two differently processed meals of similar caloric content and composition. The study will primarily focus on changes in blood cortisol levels, but other metabolic parameters will also be compared.

DETAILED DESCRIPTION:
Obesity is one of the most serious health problems of the 21st century, with ultra-processed diets being a major driver of the current obesity pandemic. Understanding how these diets affect body weight is critical to identifying new treatment targets. Current evidence suggests that the degree of food processing may affect cortisol secretion, a hormone that plays a key role in body weight regulation by increasing with acute food intake and promoting energy storage in adipose tissue. However, whether ultra-processed foods enhance cortisol response has not been thoroughly investigated.

Here, the investigators aim to understand the reaction of GCs in response to different processed foods in healthy volunteers. No medication will be used in this study.

Participants will be asked to refrain from strenuous physical activity and alcohol consumption for 24 hours prior to the study. They will fast for 12 hours before consuming a high-calorie, low-processed meal. After fasting again, participants will consume a high-calorie, ultra-processed meal on a second study day. The order of the meals is not fixed. The study will include a screening visit and two study visits.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 to 40 years
* BMI 18.5-29.9 kg/m2

Exclusion Criteria:

* Severe acute or chronic disease
* Lactose intolerance
* Severe food allergy
* Casual smoking (more than six cigarettes per day)
* Frequent, heavy alcohol consumption (more than 30g/day)
* Frequent, heavy caffeine consumption (more than 4 caffeinated drinks/day)
* Regular physical exercise (more than 4hrs per week)
* Shift work
* Previous enrollment in a clinical trial within the past two months
* Intake of any steroid-containing drugs, including topical steroids and inhalers, within four weeks of the study initiation
* Contradictions to undergo the investigated intervention
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since hormone fluctuations associated with the menstrual cycle may alter cortisol levels, women will not be included in the study. Although diversity will be reduced and the statements of the study cannot be applied to the female sex, these strict inclusion criteria allow an optimal homogeneity and increase statistical power.
Enrollment: 20 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Blood cortisol change | Up to six weeks
  Change in blood cortisol assessed by repeadidly collecting blood before and after the meal

SECONDARY OUTCOMES:
Energy expenditure (basal metabolic rate, diet-induced thermogenesis | Up to six weeks
  Basal metabolic rate measured with indirect calorimetry
Substrate utilization (respiratory quotient) | Up to six weeks
  Respiratory quotient assessed with indirect calorimetry
Body composition | Up to six weeks
  Body impedance analysis before meal
Satiety | Up to six weeks
  Appetite rating with visual analogue scale (VAS) from 0mm-100mm (0mm=not at all and 100mm=extreme)
Weight | Up to six weeks
  Measurement of weight with a standard scale
Motivation to eat | Up to six weeks
  Motivation to eat measured with a speed clicking test
Systolic and diastolic blood pressure | Up to six weeks
  Assessment of blood pressure with a standard blood pressure monitor
Lipids (total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides) | Up to six weeks
  Blood collection fasted
Perceived stress | Up to six weeks
  Measured by perceived stress questionnaire
C-peptide | Up to six weeks
  Change in blood cortisol assessed by repeadidly collecting blood before and after the meal
Insulin | Up to six weeks
  Change in blood cortisol assessed by repeadidly collecting blood before and after the meal
Blood glucose | Up to six weeks
  Change in blood glucose assessed by repeadidly collecting blood before and after the meal
Neuroendocrine hormones (thyroid hormones, GLP1, glucagon, ACTH) | Up to six weeks
  Change in blood cortisol assessed by repeadidly collecting blood before and/or after the meal

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Seelig, PD Dr. med., Principal Investigator — Sponsor and principal investigator
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No